CLINICAL TRIAL: NCT06967246
Title: Effect of Kinesio Taping of Pain, Swelling and Trismus After Mandibular Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Lam Cu Phong, lecturer, clinical professor, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UMPHCMcity
Record Dates: First submitted 2025-04-26; First posted 2025-05-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: KINESIOTAPING; Third Molar Extraction Surgery; Pain; Swelling; Trismus
MeSH Terms: conditions — Pain; Trismus | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): kinesio taping after third molar extraction on 1 side
  Interventions: Combination Product: Kinesio tape
- control group (Placebo Comparator): placebo taping after third molar extraction on the other side
  Interventions: Combination Product: non-elastic tape

INTERVENTIONS:
Combination Product: Kinesio tape — Kinesio tape applied to one surgical site
  Arms: Study group
Combination Product: non-elastic tape — The non-elastic tape with only adhesive properties was used as the placebo tape on the other side
  Arms: control group

SUMMARY:
This study evaluates the effectiveness of kinesio taping in reducing swelling, pain, and trismus complications after wisdom tooth extraction surgery. Patients undergoing bilateral symmetrical extraction of mandibular third molars, Kinesio tape was applied on the study side and placebo tape on the control side. Pain intensity was assessed using the Visual Analog Scale (VAS), swelling was measured using predefined facial landmarks, and mouth opening was recorded using interincisal distance measurements. Data were collected preoperatively (T0) and on the 1st (T1), 2nd (T2), and 3rd (T3) postoperative days.

DETAILED DESCRIPTION:
Introduction: Complications following third molar surgery can affect patients' quality of life. Kinesio taping is a simple, non-invasive method with a clear mechanism of action in fluid drainage, one of the strategies for symptom reduction in wisdom tooth extraction surgery. This study evaluates the effectiveness of kinesio taping in reducing swelling, pain, and trismus complications after wisdom tooth extraction surgery.

Methods: A split-mouth, randomized, placebo-controlled clinical trial was conducted on 17 patients indicated bilateral mandibular third molar extraction. Each patient had Kinesio tape applied to one surgical site and a placebo tape to the contralateral side. Pain intensity was assessed using the Visual Analog Scale (VAS), swelling was measured using predefined facial landmarks, and mouth opening was recorded using interincisal distance measurements. Data were collected preoperatively (T0) and on the 1st (T1), 2nd (T2), and 3rd (T3) postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Patients have bilaterally impacted mandibular third molars that are relatively symmetrical and have the same difficulty according to Pell and Gregory's classification, with an angulation difference between the two teeth not exceeding 15°. The angulation of each third molar is measured on a panoramic X-ray as the angle formed between the long axis of the third molar and the adjacent second molar.
* Patients do not have preoperative symptoms of swelling or pain.
* Patients agree to participate in the study after receiving a clear explanation and counseling.

Exclusion Criteria:

* Patients with systemic conditions contraindicating tooth extraction surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
post operative pain | 1st, 2nd, 3rd post operative days
  * Pain intensity was evaluated using the Visual Analog Scale (VAS) and the total number of analgesic tablets consumed by the patient. Patients self-assessed their pain levels using VAS during the first 3 days after surgery.
  * The VAS is a 100 mm long straight segment from 0 (painless) to 100 (unbearable pain).
post operative swelling | 1st, 2nd, 3td postoperative day
  - Preoperative facial measurements were recorded by assessing the lengths of the following segments:
  * AB (vertical dimension): From the outer canthus (A) to the lowest point of the mandibular angle (B).
  * CD line (horizontal dimension): from the midpoint of the tragus (C) to the oral commissure (D).
  * BD line (oblique dimension): from the lowest point of the mandibular angle (B) to the oral commissure (D).
  On each assessment timepoint:
  - The patient sat in a 45-degree reclined chair position with the lower jaw in the resting position. Swelling was assessed by re-measuring 3 segments: AB, CD and BD during the first 3 days after surgery.

SECONDARY OUTCOMES:
Number of painkiller tablets: | 1st, 2nd, 3rd post operative days
  record the total number of painkiller tablets taken by the patient and summarize on the 3rd day after surgery.
post operative trismus | 1st, 2nd, 3td postoperative day
  The patient's maximum mouth opening was assessed using a caliper to measure the interincisal distance, rounded to the nearest millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh city, Ho Chi Minh City, Vietnam